CLINICAL TRIAL: NCT06762249
Title: Combined Effect of Constraint Induced Movement Therapy and Brunnstrom Movement Therapy on Upper Extremity Spasticity, Motor Activity and Quality of Life in Stroke Patients
Brief Title: Combined Effect of CIMT and Brunnstrom Therapy on UE in Stroke Patients
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/24/0250
Record Dates: First submitted 2025-01-01; First posted 2025-01-07 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2025-01

CONDITIONS: Stroke Patients
Keywords: Brunnstrom movement therapy; Constraint induced movement therapy; motor activity; quality of life; spacticity; stroke patients
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CIMT+ Brunnstrom therapy + routine physical therapy. (Experimental): Group A participants will receive Constraints innduced movement therapy and Brunnstrom movement therapy along with routine physical therapy This therapy will be given as 5 days session for 4 weeks.
  Interventions: Other: CIMT + Brunnstrom therapy + routine physical therapy
- CIMT + routine physical therapy (Active Comparator): Group B participants will receive Constraint Induced movement therapy along with routine physical therapy exercises. This therapy will be given for 4 weeks.
  Interventions: Other: CIMT + routine physical therapy

INTERVENTIONS:
Other: CIMT + Brunnstrom therapy + routine physical therapy — this therapy will be given for 5 days per week for 4 weeks.
  Arms: CIMT+ Brunnstrom therapy + routine physical therapy.
Other: CIMT + routine physical therapy — this therapy will be given for 5 days per week for 4 weeks
  Arms: CIMT + routine physical therapy

SUMMARY:
Stroke is a leading cause of disability characterized by inadequate blood supply to the brain, leading to cell death and neurological deficits. Motor impairment of the upper extremity is a common consequence among stroke patients, resulting in paralysis of the upper limb. Both Constraint Induced Movement Therapy and Brunnstrom therapy have shown promise in improving motor activity and overall quality of life in stroke patients.This randomized controlled trial will be carried out at in Multan over 10 months. Total number of 56 participants meeting the inclusion criteria will be included in this study. Participants will be randomly assigned into 2 groups . Both groups will receive interventions for five days a week for 4 weeks.

DETAILED DESCRIPTION:
Stroke is the leading cause of death and disability worldwide. Remarkably, approximately 90 percent of strokes have modifiable risk factors, indicating that stroke prevention is largely possible. UE impairments are the common consequence among stroke patients, resulting in a higher likelihood of residual paralysis in the upper limb. These impairments significantly affect the performance of daily activities and diminish patients' quality of life.This study aims to determine the combined effects of constraint induced movement therapy and brunnstrom movement therapy on upper limb spasticity, motor activity and quality of life in stroke patients. This randomized controlled trial will be carried out at in Multan over 10 months after approval of synopsis. Total number of 56 participants meeting the inclusion criteria will be included in this study through a non-probability convenience sampling technique. Participants will be randomly assigned into 2 groups using computer generated method. Group A participants will receive both CIMT and brunnstrom movement therapy with routine physical therapy while Group B participants will receive only CIMT with routine physical therapy. Both groups will receive interventions for five days a week for 4 weeks. The outcome measuring sacales used will be FMUE scale to assess motor activity, FIM scale to assess spasticity and Modified Ashworth scale to assess spasticity. For within group analysis paired t-test will be applied for parametric data. For between group analysis independent t-test will be applied for parametric data. Data analysis will be performed by using SPSS 28 version.

ELIGIBILITY:
Inclusion Criteria:

* Age group between 40 and 70 years
* Both male and female
* Patient being diagnosed with hemiplegic stroke
* Patient having hemorrhagic stroke or ischemic stroke
* Patient able to give their consent for rehabilitation program
* Patient having 24 or higher score from Standardized Mini-Mental Test
* Patient being able to stand for 2 min without assistance from a person

Exclusion Criteria:

* Patient with cognitive impairment or dementia
* Patient having any other disease that prevents participation in the rehabilitation program
* Patient that participated in any ongoing rehabilitation program
* Patient having pain in UE 4 or higher according to the Visual Analog Scale which is scored 0-10
* Patient had spasticity in any joint of the UE and scored 2 or higher according to the Modified Ashworth Scale

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-02-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
Fugl-Meyer Upper Extremity Motor Evaluation Scale (FM-UE) | 4 weeks
  The FMA-UE consists of 30 items assessing motor function and 3 items assessing reflex function. The score most applicable to task performance is given from "0, inability," "1, beginning ability," to "2, normal"
Functional Independence Measure (FIM) | 4 weeks
  The scale consists of six sub-headings and a total of 18 items. Scores that can be obtained from the scale range from 18-126, and higher scores indicate that the individual is more independent in daily life
Modified Ashworth scale | 4 weeks
  The modified Ashworth scale is a muscle tone assessment scale used to assess the resistance experienced during passive range of motion, which does not require any instrumentation and is quick to perform.
Mini Mental state examination | 4 weeks
  The MMSE is a widely used cognition screening test. It has a maximum score of 30 points. It assesses aspects of orientation, recall, language and visual construction.

CONTACTS AND LOCATIONS:
Overall Officials: Sabiha Arshad, Principal Investigator — Riphah International University
Locations (2):
- Pakistan (2):
  - Azeem Electroneurophysiology diognostic and Physiotherapy center Multan, Multan, Punjab Province
  - Qaisrani Hospital Multan, Multan, Punjab Province

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abba M, Muhammad A, Badaru U, Abdullahi A. Comparative effect of constraintinduced movement therapy and proprioceptive neuromuscular facilitation on upper limb function of chronic stroke survivors. Physiotherapy Quarterly. 2020;28(1):1-5.
- [Background] . Shaheen S, Afzal B, Tahir M, Mahmood U, Yousaf F, Tariq F. Combined Effects of Brunnstorm Movement Therapy and Low-Level Laser Therapy on Upper Limb Function and Hand Dexterity in Chronic Stroke Patient. Journal of Health and Rehabilitation Research. 2024;4(1):1457-62
- [Background] Rocha LSO, Gama GCB, Rocha RSB, Rocha LB, Dias CP, Santos LLS, Santos MCS, Montebelo MIL, Teodori RM. Constraint Induced Movement Therapy Increases Functionality and Quality of Life after Stroke. J Stroke Cerebrovasc Dis. 2021 Jun;30(6):105774. doi: 10.1016/j.jstrokecerebrovasdis.2021.105774. Epub 2021 Apr 10. PMID 33848906
- [Background] Terranova TT, Simis M, Santos ACA, Alfieri FM, Imamura M, Fregni F, Battistella LR. Robot-Assisted Therapy and Constraint-Induced Movement Therapy for Motor Recovery in Stroke: Results From a Randomized Clinical Trial. Front Neurorobot. 2021 Jul 21;15:684019. doi: 10.3389/fnbot.2021.684019. eCollection 2021. PMID 34366819
- [Background] Nasb M, Li Z, S A Youssef A, Dayoub L, Chen H. Comparison of the effects of modified constraint-induced movement therapy and intensive conventional therapy with a botulinum-a toxin injection on upper limb motor function recovery in patients with stroke. Libyan J Med. 2019 Dec;14(1):1609304. doi: 10.1080/19932820.2019.1609304. PMID 31032717
- [Background] Puri S, Kovela RK, Qureshi MI, Dadgal R, Timothy R, Samal S. Effect of Brunnstrom Movement Therapy Combined with Neurodevelopmental Therapy on Balance and Mobility in a Patient with Acute Stroke: An Interesting Case Report. JPRI. 2022:6-9.
- [Background] Dhanalakshmi L, Alagesan J, Buvanesh A. Effectiveness of Constraint Induced Movement Therapy and Proprioceptive Neuromuscular Facilitation on Upper Extremity Functions in Stroke. Indian Journal of Physiotherapy & Occupational Therapy. 2024;18.
- [Background] Akter R, Sharma N, Ahmed S, Srivastav AK. Combined effect of Brunnstrom's hand rehabilitation and functional electrical stimulation for improving hand function in patients with chronic stroke: A randomized controlled trial. J Bodyw Mov Ther. 2023 Jul;35:84-90. doi: 10.1016/j.jbmt.2023.04.021. Epub 2023 Apr 28. PMID 37330808